CLINICAL TRIAL: NCT06188689
Title: Evaluation of a Clinical Diagnostic Test for Calcium Release Deficiency Syndrome: The DIAGNOSE CRDS Study
Brief Title: Evaluation of A Clinical Diagnostic Test for CRDS
Acronym: DIAGNOSE CRDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14546
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Calcium Release Deficiency Syndrome (CRDS)
Keywords: cardiac arrhythmia, sudden cardiac death, cardiac ryanodine receptor, unexplained cardiac arrest
MeSH Terms: conditions — Arrhythmias, Cardiac; Death, Sudden, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pacing (Experimental): Separate ventricular and atrial pacing trains will be administered at different cycle lengths and the ventricular repolarization response on the first sinus beat following the subsequent pause will be evaluated.
  Interventions: Diagnostic Test: Pacing

INTERVENTIONS:
Diagnostic Test: Pacing — 1. Ventricular 10 beat burst at 500ms (120bpm)
  2. Ventricular 10 beat burst at 400ms (150bpm)
  3. Atrial 10 beat burst at 500ms (120bpm)
  4. Atrial 10 beat burst at 400ms (150bpm).

SUMMARY:
Calcium Release Deficiency Syndrome (CRDS) is a novel inherited arrhythmia syndrome secondary to RyR2 loss-of-function that confers a risk of sudden cardiac death. Diagnosis of CRDS presently requires cellular-based in vitro confirmation that an RyR2 variant causes loss-of-function. We hypothesize that CRDS can be diagnosed clinically through evaluation of the repolarization response to brief tachycardia, mediated by cardiac pacing, and a subsequent pause.

DETAILED DESCRIPTION:
RyR2 loss-of-function variants have recently been established as causative for a new disease termed calcium release deficiency syndrome (CRDS) that confers a risk of malignant ventricular arrhythmias and sudden cardiac death. RyR2 encodes the cardiac ryanodine receptor, the calcium release channel on the sarcoplasmic reticulum that mediates excitation-contraction coupling through calcium-induced calcium-release. In contrast to CRDS, pathogenic RyR2 gain-of-function variants result in an autosomal dominant form of catecholaminergic polymorphic ventricular tachycardia (CPVT). The adrenergic-mediated ventricular arrhythmias characteristic of CPVT can be readily reproduced on exercise stress testing (EST), making EST the standard clinical diagnostic tool for CPVT.

In contrast to CPVT, the CRDS clinical phenotype is concealed with standard cardiac testing tools and its diagnosis presently requires cellular-based in vitro confirmation that an RyR2 variant causes loss-of-function. Beyond the significant time delay associated with in vitro functional analysis, this testing requires specialized expertise that is not widely available and remains research-based, making it impractical for routine use in clinical care. In this overall context, it is likely that the vast majority of global CRDS cases have yet to be diagnosed.

A prior report of an "atypical CPVT" family carrying an RyR2-p.M4109R variant observed marked and transient repolarization changes following pacing mediated tachycardia and a subsequent pause. Since publication of this report, in vitro characterization of the RyR2-p.M4109R variant has confirmed its being loss-of-function and the familial diagnosis has been revised to CRDS. Driven by these observations and promising preliminary findings, the DIAGNOSE CRDS study seeks to further investigate this apparent electrocardiographic signature of CRDS following brief tachycardia and subsequent pause as a potential method to clinically diagnose the condition.

ELIGIBILITY:
Cohort 1: Calcium Release Deficiency Syndrome (CRDS) Cases

Inclusion criteria:

• Presence of an RyR2 variant confirmed to be loss-of-function on in vitro testing

Exclusion criteria:

• Unable to provide informed consent

Cohort 2: Catecholaminergic Polymorphic Ventricular Tachycardia (CPVT) Cases

Inclusion criteria:

* Satisfy a clinical phenotype consistent with the Expert Consensus Statement
* Presence of a confirmed or presumed pathogenic gain-of-function RyR2 variant OR homozygous or compound heterozygous for likely pathogenic/pathogenic CASQ2 variants

Exclusion criteria:

* Unable to provide informed consent
* Use of a QT prolonging medication, aside from flecainide, at the time of the burst pacing maneuvers

Cohort 3: Survivors of Unexplained Cardiac Arrest (UCA)

Inclusion criteria:

* Cardiac arrest requiring cardioversion or defibrillation that remains unexplained following an ECG, echocardiogram, coronary assessment, cardiac MRI, and exercise treadmill test
* Undergone genetic testing that includes screening of RyR2*

Exclusion criteria:

* Unable to provide informed consent
* Use of a QT prolonging medication at the time of the burst pacing maneuvers

  * Among survivors of UCA that possess a rare RyR2 variant in the absence of a CPVT phenotype, in vitro functional testing will be performed in order to confirm it is not loss- or gain-of-function (and will be arranged through the laboratory of Dr. Wayne Chen at the University of Calgary).

Cohort 4: SVT controls

Inclusion criteria:

• Undergoing an invasive electrophysiology study

Exclusion criteria:

* Ventricular cardiomyopathy
* Ventricular pre-excitation
* Long QT syndrome
* Use of a QT prolonging medication at the time of the EP study
* Use of a Class I or Class III anti-arrhythmic drug at the time of the EP study
* Known obstructive coronary artery disease (existing coronary stenosis >50%)
* Unable to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
ΔT-wave amplitude value | At time of pacing maneuver
  T-wave amplitude on first post-pause sinus beat subtracted by the T-wave amplitude on the last sinus beat prior to pacing
ΔQT value | At time of pacing maneuver
  Absolute QT value on first post-pause sinus beat subtracted by the absolute QT value on the last sinus beat prior to pacing

SECONDARY OUTCOMES:
Absolute QT value | At time of pacing maneuver
  Absolute QT value on first post-pause sinus beat
Absolute T-wave amplitude | At time of pacing maneuver
  Absolute T-wave amplitude on first post-pause sinus beat

CONTACTS AND LOCATIONS:
Overall Officials: Ziv Dadon, MD, Study Director — Shaare Zedek Medical Center; Jason D Roberts, MD MAS, Principal Investigator — McMaster University; Wayne Chen, PhD, Principal Investigator — University of Calgary
Locations (18):
- United States (3):
  - University of California, San Francisco, California
  - Mayo Clinic, Rochester, Minnesota
  - University of Washington, Seattle, Washington
- Belgium (2):
  - Antwerp University Hospital, Edegem, Antwerp
  - Universitair Ziekenhuis Brussel, Brussels
- Canada (9):
  - University of Calgary, Calgary, Alberta
  - Children's & Women's Health Centre of British Columbia, Vancouver, British Columbia
  - The University of British Columbia, Vancouver, British Columbia
  - Hamilton General Hospital, Hamilton, Ontario
  - London Health Sciences Centre - University Hospital, London, Ontario
  - Ottawa Heart Institute, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Montréal Heart Institute, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec-Université Laval, Québec, Quebec
- Aarhus University Hospital, Aarhus, Denmark
- CHU de Bordeaux, Bordeaux, Nouvelle-Aquitaine, France
- Shaare Zedek Medical Center, Jerusalem, Israel
- Oxford University Hospitals, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sun B, Yao J, Ni M, Wei J, Zhong X, Guo W, Zhang L, Wang R, Belke D, Chen YX, Lieve KVV, Broendberg AK, Roston TM, Blankoff I, Kammeraad JA, von Alvensleben JC, Lazarte J, Vallmitjana A, Bohne LJ, Rose RA, Benitez R, Hove-Madsen L, Napolitano C, Hegele RA, Fill M, Sanatani S, Wilde AAM, Roberts JD, Priori SG, Jensen HK, Chen SRW. Cardiac ryanodine receptor calcium release deficiency syndrome. Sci Transl Med. 2021 Feb 3;13(579):eaba7287. doi: 10.1126/scitranslmed.aba7287. PMID 33536282
- [Result] Nof E, Belhassen B, Arad M, Bhuiyan ZA, Antzelevitch C, Rosso R, Fogelman R, Luria D, El-Ani D, Mannens MM, Viskin S, Eldar M, Wilde AA, Glikson M. Postpacing abnormal repolarization in catecholaminergic polymorphic ventricular tachycardia associated with a mutation in the cardiac ryanodine receptor gene. Heart Rhythm. 2011 Oct;8(10):1546-52. doi: 10.1016/j.hrthm.2011.05.016. Epub 2011 May 26. PMID 21699856
- [Result] Ormerod JOM, Ormondroyd E, Li Y, Taylor J, Wei J, Guo W, Wang R, Sarton CNS, McGuire K, Dreau HMP, Taylor JC, Ginks MR, Rajappan K, Chen SRW, Watkins H. Provocation Testing and Therapeutic Response in a Newly Described Channelopathy: RyR2 Calcium Release Deficiency Syndrome. Circ Genom Precis Med. 2022 Feb;15(1):e003589. doi: 10.1161/CIRCGEN.121.003589. Epub 2021 Dec 24. PMID 34949103
- [Result] Roston TM, Wei J, Guo W, Li Y, Zhong X, Wang R, Estillore JP, Peltenburg PJ, Noguer FRI, Till J, Eckhardt LL, Orland KM, Hamilton R, LaPage MJ, Krahn AD, Tadros R, Vinocur JM, Kallas D, Franciosi S, Roberts JD, Wilde AAM, Jensen HK, Sanatani S, Chen SRW. Clinical and Functional Characterization of Ryanodine Receptor 2 Variants Implicated in Calcium-Release Deficiency Syndrome. JAMA Cardiol. 2022 Jan 1;7(1):84-92. doi: 10.1001/jamacardio.2021.4458. PMID 34730774
- [Derived] Ni M, Dadon Z, Ormerod JOM, Saenen J, Hoeksema WF, Antiperovitch P, Tadros R, Christiansen MK, Steinberg C, Arnaud M, Tian S, Sun B, Estillore JP, Wang R, Khan HR, Roston TM, Mazzanti A, Giudicessi JR, Siontis KC, Alak A, Acosta JG, Divakara Menon SM, Tan NS, van der Werf C, Nazer B, Vivekanantham H, Pandya T, Cunningham J, Gula LJ, Wong JA, Amit G, Scheinman MM, Krahn AD, Ackerman MJ, Priori SG, Gollob MH, Healey JS, Sacher F, Nof E, Glikson M, Wilde AAM, Watkins H, Jensen HK, Postema PG, Belhassen B, Chen SRW, Roberts JD. A Clinical Diagnostic Test for Calcium Release Deficiency Syndrome. JAMA. 2024 Jul 16;332(3):204-213. doi: 10.1001/jama.2024.8599. PMID 38900490